CLINICAL TRIAL: NCT04646928
Title: Efficacy of Entecavir for Reducing the Risk of Hepatocellular Carcinoma in Chronic Hepatitis B Patients With Compensated Cirrhosis and Low Viral Load: a Multicenter, Prospective Study
Brief Title: Study of Entecavir for Reducing the Risk of Hepatocellular Carcinoma in Chronic Hepatitis B Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHA University (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EN-REACH
Record Dates: First submitted 2020-11-22; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hepatitis B virus (HBV) DNA level from patient blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
To analyze the incidence of liver cancer after entecavir administration among patients with low viral load and cirrhosis due to chronic hepatitis B infection.

DETAILED DESCRIPTION:
To analyze the incidence of liver cancer after entecavir administration among patients with low viral load (HBV DNA titer<2,000 IU/mL (104 copies/mL)) and cirrhosis due to chronic hepatitis B infection.

ELIGIBILITY:
Inclusion Criteria:

* A subject who has consented to participate in this clinical trial
* A subject aged between ≥20 to ≤75 years old
* A subject with positive HBsAg for more than 24 weeks (may be confirmed by medical history)
* HBV DNA ≥26 IU/mL or ≤ 2,000 IU/mL at the time of screening
* A subject diagnosed with cirrhosis with one of the following:

  1. Subject with confirmed liver cirrhosis in the screening period or liver biopsy performed within 1 year from the time of screening (METAVIR score> 3, ISHAK score> 4)
  2. Two or more confirmed typical findings suggesting liver cirrhosis from imaging such as liver ultrasound and CT performed within 24 weeks of screening or during screening period (nodularity of the liver surface, atrophy of the inner right and left lobes, thickening of the left and tail lobes, hepatic portal system expansion of surrounding space, expansion of hepatic portal system (>1.3 cm) and splenomegaly (>12 cm))
  3. One or more confirmed typical findings suggesting liver cirrhosis from imaging such as liver ultrasound and CT performed within 24 weeks of screening or during screening period (nodularity of the liver surface, atrophy of the inner right and left lobes, thickening of the left and tail lobes, hepatic portal system expansion of surrounding space, expansion of hepatic portal system (>1.3 cm) and splenomegaly (>12 cm)) or findings including the following:
* Confirmed thrombocytopenia (<150,000/mm3) at the screening period or blood tests conducted within 24 weeks from the time of screening
* Confirmed identification of esophageal varicose veins or gastric varicose veins by endoscopy or CT performed within one year from the screening period or at screening
* Liver stiffness measurement (LSM)> 11.5 kilopascal (kPa) (F4) as a result of liver fibrosis scan, performed within 1 year from screening period or at screening

Exclusion Criteria:

* A subject with non compensated cirrhosis and any of the following:

  1. Serum bilirubin> 3 mg/dL
  2. Prothrombin time> 6 seconds prolonged or International Normalized Ratio (INR) >1.6
  3. Serum albumin <2.8 g/dL
  4. History of ascites, varicose bleeding, hepatorenal syndrome, hepatic encephalopathy (hepatic coma) requiring treatment within 5 years from screening
  5. Child-Pugh score ≥ 8
* A subject who have received interferon or other oral nucleic acid analogues (nucleos(t)ide analogues) (However, if the treatment duration was less than 30 days in the past and the treatment was treated 24 weeks before the screening, participation is possible)
* A subject diagnosed with liver cancer in the past or present
* Renal function decline (creatinine clearance <50 mL/min, estimated by the Cockcroft-Gault formula)
* A subject with serious concomitant diseases such as congestive heart failure, chronic kidney disease, blood disease, or malignant tumors in the past or present
* A subject infected with hepatitis C virus (HCV) or human immunodeficiency virus (HIV)
* A subject who consume excessive alcohol (men: 30g/day or more, women: 20g/day or more)
* A subject with liver diseases such as autoimmune hepatitis, hemochromatosis, or Wilson's disease
* Pregnant or breastfeeding women
* Previous organ transplant recipients
* A subject unable to complete the clinical trial or to have any medical condition that may interfere with the evaluation of the efficacy of this clinical trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with Hepatitis B and liver cirrhosis displaying low viral load (HBV DNA titer <2,000 IU/mL (104 copies/mL))
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2022-05-28 (Estimated); Study Completion 2022-08-26 (Estimated)

PRIMARY OUTCOMES:
5-year Cumulative hepatocellular carcinoma incidence | 5 years
  Compare the difference in the 5-year cumulative incidence of hepatocellular carcinoma in patients with chronic hepatitis B and cirrhosis with entecavir and control

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Compare the difference in the 5-year incidence overall survival in patients with chronic hepatitis B and cirrhosis with entecavir and control
Incidence of ascites, esophageal, gastric variceal bleeding, hepatic encephalopathy (hepatic coma) | 5 years
  Compare the difference in the 5-year incidence of ascites/esophageal/gastric variceal bleeding/hepatic encephalopathy (hepatic coma) in patients with chronic hepatitis B and cirrhosis with entecavir and control
Incidence of virologic response, virologic breakthrough | 5 years
  Compare the difference in the 5-year incidence incidence of virologic response and virologic breakthrough in patients with chronic hepatitis B and cirrhosis with entecavir and control
Incidence of cirrhosis regression | 5 years
  Compare the difference in the 5-year incidence of cirrhosis regression in patients with chronic hepatitis B and cirrhosis with entecavir and control

CONTACTS AND LOCATIONS:
Overall Officials: SungKyu Hwang, MD, Principal Investigator — Principal Investigator
Locations (11):
- South Korea (11):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Bundang Jesaeng Hospital, Gyeonggi-do
  - Catholic University of Korea, Uijeongbu ST. Mary's Hospital, Gyeonggi-do
  - CHA Bundang Medical Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Gachon University, Donginchoen Gil Hospital, Sŏngnam
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon